CLINICAL TRIAL: NCT02878447
Title: The Utility of External Beam Radiotherapy for Haemoptysis Secondary to Aspergillomata and Structural Lung Diseases in Patients Who Are Refractory to Medical Management and Not Surgical Candidates: A Pilot Study
Brief Title: The Utility of Radiotherapy in the Management of Haemoptysis Secondary to Aspergillomata and Structural Lung Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Stellenbosch (Other)
Responsible Party: Principal Investigator, Dr Brian Allwood, Principal investigator, University of Stellenbosch
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M15/09/033
Record Dates: First submitted 2016-06-23; First posted 2016-08-25 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Haemoptysis
Keywords: Haemoptysis; Radiotherapy; Tuberculosis; Aspergilloma; Bronchiectasis
MeSH Terms: conditions — Hemoptysis; Tuberculosis; Bronchiectasis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- External Beam Radiotherapy (Experimental): Patients will receive radiotherapy (3.5Gy weekly for 5 fractions to a maximum of 17G) prescribed to a central plane using mega-voltage radiation encompassing all the assessed affected lung tissue
  Interventions: Radiation: External beam radiotherapy
- Control (No Intervention): Patients will receive best medical care.

INTERVENTIONS:
Radiation: External beam radiotherapy — External beam radiotherapy will be prescribed to a central plane using mega-voltage radiation encompassing all the assessed affected lung tissue at 3.5Gy weekly for 5 fractions to a maximum of 17G
  Arms: External Beam Radiotherapy

SUMMARY:
The sequelae of tuberculosis are still the commonest causes of haemoptysis in the developing world, where life-threatening haemoptysis remains a common and not infrequently fatal medical emergency. Haemoptysis can be life-threatening either as a result of compromised gas exchange or because of circulatory collapse secondary to acute blood loss. Haemodynamic and ventilatory support, followed by bronchial artery embolisation (BAE) as a bridge to potentially curative treatment such as lung resection, remains the standard of care. Often patients do not qualify for surgical intervention and BAE is, at best, a temporary solution. External beam radiotherapy (EBRT) may be an alternative, curative intervention in the management of haemoptysis in patients with no alternative options. There is a paucity of studies reporting the use of EBRT in patients without malignancy and with regards to specific doses of EBRT. This pilot study aims to explore the potential of varying doses of EBRT in the management of massive haemoptysis.

DETAILED DESCRIPTION:
Currently the best curative treatment of massive haemoptysis is surgical resection of the affected portion of lung. For patients who do not qualify for surgery, there are few alternative interventions, most of which only provide a temporary solution.

Surgical resection of the diseased areas, which offers the possibility of cure, is best performed as an elective procedure. It carries a not insignificant mortality, with reports varying between 1% and 50%. Unfortunately, many patients admitted to Tygerberg Academic Hospital, are not candidates for either elective or emergency surgical resection. The most common reasons for inoperability are: irresectable disease (i.e. damage to the lungs is bilateral and too extensive to allow resection, or the site of bleeding is not known); or severely reduced cardiopulmonary reserves secondary to extensive pre-existing lung damage, making lung resection surgery impossible due to excessively high mortality risk.

Repeat BAE (as a palliative measure in inoperable cases) is not always technically feasible and does not always lead to cessation of the bleeding. Additionally long term recurrence rates following BAE are variable estimated at between 18-42%, and carries a high mortality.

A significant number of patients with massive haemoptysis do not qualify for either surgery or BAE, thus rendering them without treatment option, save palliation with long-term opiates. Their fate is that of recurrent haemoptysis and a high associated mortality. Endobronchial occluding devices have been considered, however their high cost and required expertise prohibits their extensive use.

A novel treatment of this condition potentially is external beam radiotherapy (EBRT). A case report of five patients has documented EBRT in the setting of mycetoma where between 7 and 14Gy was used, with cessation of life threatening haemoptysis. However follow-up was limited to 6 months, and the effects of EBRT in the setting of post-tuberculous structural lung disease without mycetoma is not known. The potential mechanism of the achieved haemostasis was speculated as being the induction of radiation damage to the radiosensitive capillaries, with subsequent inflammatory response, in keeping with previous rat models of lung perfusion following high dose (30Gy) EBRT exposure.

There is therefore a paucity of data on the utility of EBRT in benign conditions such bronchiectasis and aspergillomata. Furthermore due to the different effects, particularly temporal, the radiation has on normal and benign conditions it is difficult to extrapolate from the malignant scenario to the benign. Laboratory studies have however demonstrated the effects of high dose radiation on tissue that may result in a reduced bleeding tendency.

This study aims to explore a novel therapeutic strategy for patients with life-threatening haemoptysis who are not candidates for definitive management (i.e. lung resection). This study also aims to establish if there is a measurable response to varying doses of chest radiation in cases of haemoptysis caused by benign conditions.

This study is a prospective randomised control-intervention study. Patients will be allocated to one of 2 arms (control and EBRT at 3.5Gy weekly for 5 fractions to a maximum of 17G). The primary outcome will be time to recurrent haemoptysis. Secondary outcomes include physical performance, lung function and the occurrence of EBRT complications. Patients will be followed up daily whilst in hospital and for one year post intervention.

Assessors and those performing the statistical analysis will be blinded to the group allocation. Statistical analysis will include univariate and multivariate analysis with appropriate parametric or non-parametric tests. Appropriate tests for categorical data (e.g. Chi-squared test) and continuous data (e.g. Kruskal-Wallis, and ANOVA) will be used. Logistic and linear regression modelling will be used for certain outcomes, and multivariate analysis will be performed using step-wise regression modelling and full modelling where appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects, 18 years of age and older.
* Written informed consent provided by patient
* Current or previously documented admission to hospital with large volume haemoptysis (>200ml); or haemoptysis with haemodynamic compromise (SBP < 100mmHg for 15 minutes) or requiring fluid resuscitation; haemoptysis requiring intubation or deemed life-threatening by attending clinicians.
* The cause of haemoptysis must be due to severe underlying lung destruction/ bronchiectasis, post-tuberculous lung damage or the presence of an aspergillomata.
* Primary bronchial artery embolisation not considered technically possible or failed BAE
* Lung resection not possible because of poor cardiopulmonary reserves (as defined by the current ERS/ESTS clinical guidelines, independently reviewed by a team of consisting of a thoracic surgeon, pulmonologist and anaesthetist who will need to be in agreement on inoperability and/or lack of cardiopulmonary reserve)

Exclusion Criteria:

* Active tuberculosis
* High clinical suspicion of lung carcinoma
* Known deep venous thrombosis or pulmonary embolism
* Any social or psychological condition that may impair insight or compliance with the study including follow up
* Any other condition, which in the opinion of the investigators, places the subject at increased risk for transport and administration of EBRT e.g. severe haemodynamic instability, mechanical ventilation with high FiO2 requirements etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Composite end-point of time to recurrent life-threatening haemoptysis, or death | 1 year

SECONDARY OUTCOMES:
Six minute walk test | 1 year
  Improvement from baseline
Time to massive haemoptysis (>200mL per day) | 1 year
Fev1/FVC | 1 year
  Improvement from baseline
Total lung capacity (TLC) Total lung capacity (TLC) | 1 year
  Improvement from baseline
Diffusion capacity (DLCO) Total lung capacity (TLC) | 1 year
  Improvement from baseline
Radiological change in volume (maximum diameters in three planes) | 1 year
  Performed by two radiologists to determine the radiological resolution of aspergillomata
Number of complications associated with Radiotherapy | 1 year
  nausea, skin changes, pulmonary infection, pain etc.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Allwood, MBChB, PhD, Study Chair — University of Stellenbosch
Locations (1):
- University of Stellenbosch, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fernando HC, Stein M, Benfield JR, Link DP. Role of bronchial artery embolization in the management of hemoptysis. Arch Surg. 1998 Aug;133(8):862-6. doi: 10.1001/archsurg.133.8.862. PMID 9711960
- [Background] von Groote-Bidlingmaier F, Koegelenberg CF, Bolliger CT. Functional evaluation before lung resection. Clin Chest Med. 2011 Dec;32(4):773-82. doi: 10.1016/j.ccm.2011.08.001. PMID 22054885
- [Background] Brunelli A, Charloux A, Bolliger CT, Rocco G, Sculier JP, Varela G, Licker M, Ferguson MK, Faivre-Finn C, Huber RM, Clini EM, Win T, De Ruysscher D, Goldman L; European Respiratory Society and European Society of Thoracic Surgeons joint task force on fitness for radical therapy. ERS/ESTS clinical guidelines on fitness for radical therapy in lung cancer patients (surgery and chemo-radiotherapy). Eur Respir J. 2009 Jul;34(1):17-41. doi: 10.1183/09031936.00184308. PMID 19567600
- [Background] Koegelenberg CF, Bruwer JW, Bolliger CT. Endobronchial valves in the management of recurrent haemoptysis. Respiration. 2014;87(1):84-8. doi: 10.1159/000355198. Epub 2013 Dec 4. PMID 24334859
- [Background] Falkson C, Sur R, Pacella J. External beam radiotherapy: a treatment option for massive haemoptysis caused by mycetoma. Clin Oncol (R Coll Radiol). 2002 Jun;14(3):233-5. doi: 10.1053/clon.2002.0063. PMID 12109828